CLINICAL TRIAL: NCT00129155
Title: Unrelated Reduced Intensity Conditioning With Treosulfan® for Allogeneic Stem Cell Transplantation in Patients With Hematological Malignancies
Brief Title: MiniMUD Study - Unrelated Reduced Intensity Conditioning With Treosulfan® for Allogeneic Stem Cell Transplantation in Patients With Hematological Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003.332
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Hematological Malignancies; Allogeneic Transplantation
Keywords: Allogenic stem cell transplantation; Treosulfan; Haematological malignancies; allogeneic stem cell transplantation in patients with hematological malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — treosulfan

INTERVENTIONS:
Drug: treosulfan

SUMMARY:
In this study, treosulfan is evaluated for conditioning in allogenic stem cell transplantation. The procedure and the follow-up are the same as in standard allogenic transplant.

The donor is unrelated (identical HLA). The graft is haematological peripheral blood stem cell.

The conditioning with reduced intensity is: fludarabine (from day -6 to day -2), treosulfan (from day -6 to day -4) and thymoglobuline (from day -2 to day -1).

ELIGIBILITY:
Inclusion Criteria:

* AGE: >= 18 years and <= 65 years
* Patients with a too high transplant-related mortality (TRM) after standard transplantation (multiple myeloma, chronic lymphoid leukemia, non Hodgkin's lymphoma, myelodysplasia)
* Patients with visceral contra-indication for standard transplantation:

  * cardiac: myocardiopathy; forced expiratory volume (FEV) < 50%;
  * respiratory: abnormal carbon monoxide diffusing capacity (DLCO);
  * renal: creatinine clearance < 50ml/min;
  * hepatic: transaminases and bilirubin > 2 upper normal limit;
  * infectious: controlled fungal infection.
* Karnofsky score >= 70%
* Unrelated donor HLA identical (ABC, DRB1; DQB1)
* Signed informed consent

Diagnosis :

Chronic myelogenous leukemia (CML):

* In first chronic phase, resistant to interferon with or without aracytine or refractory or resistant to Glivec
* In complete response (CR) or in 2nd partial response (PR) after being in blastic phase

Multiple myeloma (MM):

* Relapse after autograft if the therapeutic response was evaluated to 50%

Non-Hodgkin's lymphoma (NHL):

* Mantle cell lymphoma after first relapse but in case of chemosensitivity ≥ 50% except for high grade lymphoma
* In 2nd CR or PR chemosensitive in response ≥ 50% after autograft

Chronic lymphocytic leukemia (CLL):

* In 2nd CR or PR or in response ≥ 50% after autograft or in 2nd relapse after 2 lines of treatment but in case of chemosensitivity ≥ 50%

Acute myeloid leukemia (AML):

* In 2nd CR or in 1st CR for high risk criteria [high risk criteria defined by: LAM 7; leukocytes > 30,000/mm3; chromosomal abnormalities: t(6,9); abnormalities of 11q23, 17p, 11q, 20q, 21q, -5, del(5q), -7/del7q, del 9q et inv 3q]

Acute lymphoblastic leukemia (ALL):

* In 2nd CR or in 1st CR if high risk criteria patients who are defined by chromosomal abnormalities t(9,22); t(1,19); t(4,11); abnormalities of 11q23

Myelodysplastic syndromes (MDS):

* Patients without prior chemotherapy, with intermediate or high International Prognostic Scoring System (IPSS) score and blast cells < 1% in bone marrow (BM)
* CR or PR after chemotherapy for patients with 20 to 30% of blast cells in BM
* Secondary AML patients with a response to chemotherapy (< 30% blasts in BM and < 5% of blast cells in blood)

For all:

* Adequate contraception in female patients of child bearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-02

PRIMARY OUTCOMES:
Overall survival at 1 year

SECONDARY OUTCOMES:
Engraftment evaluation
Acute and chronic graft-versus-host disease incidence and severity
Response rate and survival without progression
Evaluation of conditioning and transplant toxicity
Chimerism evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Mauricette MICHALLET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot, Lyon, France